CLINICAL TRIAL: NCT00281996
Title: Phase I/II Study of Gleevec (Imatinib Mesylate, Formerly Known as STI571) and Gemcitabine for Advanced Pancreas Cancer
Brief Title: Imatinib Mesylate and Gemcitabine in Treating Patients With Locally Advanced, Metastatic, or Recurrent Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed to accrual to allow enrollment on another more promising trial.
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 02I8; NU-02I8; NU-0948-003
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine — Administered intravenously over 30 minutes on days 1 and 8 of a 21-day cycle starting at a dose of 700 mg/m2 and increasing to 1000mg/m2 by cohorts
Drug: Imatinib mesylate — Administered orally once daily with 8 ounces of water at a starting dose of 300 mg/day and increased to 600 mg/day according to cohort.
  Other Names: Gleevec

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving imatinib mesylate together with gemcitabine may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving imatinib mesylate together with gemcitabine and to see how well they work in treating patients with locally advanced, metastatic, or recurrent pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of imatinib mesylate and gemcitabine hydrochloride in patients with locally advanced, metastatic, or recurrent pancreatic cancer.
* Determine the clinical response rate in patients treated with this regimen.
* Determine the 6-month and overall survival of patients treated with this regimen.

Secondary

* Determine the toxicity profile of this regimen in these patients.
* Correlate response with expression of platelet-derived growth factor (PDGF) and PDGF receptor in tumor tissue from patients treated with this regimen.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

* Phase I: Patients receive oral imatinib mesylate once daily on days 1-14 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8*. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-5 patients receive escalating doses of imatinib mesylate and gemcitabine hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 5 or 3 of 5 patients experience dose-limiting toxicity.

NOTE: *The first cohort receives gemcitabine hydrochloride on days 1, 8, and 15

* Phase II: Patients receive imatinib mesylate and gemcitabine hydrochloride at the MTD determined in phase I in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed pancreatic cancer

  * Locally advanced, metastatic, or recurrent disease
* Measurable or evaluable disease by physical exam, plain radiographs, CT scan, or MRI
* No brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy of 12 weeks or greater
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* No chronic liver disease (i.e., chronic active hepatitis or cirrhosis)
* Creatinine ≤ 2.0 mg/dL
* No chronic renal disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier-method contraception during and for ≥ 3 months after completion of study treatment
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No uncontrolled diabetes
* No active uncontrolled infection
* No other severe and/or uncontrolled medical disease
* HIV negative

PRIOR CONCURRENT THERAPY:

* No prior therapy for metastatic disease

  * Prior fluorouracil as a radiosensitizer for adjuvant therapy after surgery or for locally advanced disease is permitted if local disease has recurred or progressed ≥ 3 months after completion of therapy or disease is present outside the radiation field
* At least 2 weeks since prior major surgery
* No concurrent grapefruit or grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose according to toxicity | After 1 cycle of therapy (1 cycle = 21 days)
Clinical response rate | After every 2 cycles of study therapy (1 cycle = 21 days)
Overall survival at 6 months | After 6 months of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mary Mulcahy, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States